CLINICAL TRIAL: NCT05518006
Title: An Exploratory Investigation of Dietary Supplementation and the Effect on the Regularity of Menstrual Cycles, Hormone Balance, and Common PMS Symptoms in Females
Brief Title: An Investigation of Premama Balance and Its Effects on Hormonal Imbalances
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Sponsor funding
Sponsor: Premama Inc. (Industry)
Collaborators: Citruslabs (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 20223
Record Dates: First submitted 2022-08-24; First posted 2022-08-26 (Actual); Last update posted 2024-04-03 (Actual); Status verified 2024-04

CONDITIONS: PMS; Menstrual Discomfort; Hormone Disturbance; Menstrual Pain; Menstrual Irregularity
Keywords: PMS; Menstrual Discomfort; Hormone Disturbance; Menstrual Pain; Menstrual Irregularity
MeSH Terms: conditions — Endocrine System Diseases; Dysmenorrhea; Menstruation Disturbances

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PreMama Balance (Experimental): Each day, the participants will take 1 packet of Premama Balance, dissolved in one glass (8oz+) of water. Premama Balance may be taken with or without food. Should participants present themselves with a sensitive stomach, it is recommended to take the drink with or after a meal to avoid an upset stomach. Participants will repeat this process daily for 6 months/24 weeks (study period) until the study is complete.
  At week 12 and in week 24, the participants will take a survey and a hormone test to track progress. In total there will be 3 surveys and 3 hormone tests. Additionally, participants will fill out a weekly consumption survey to track compliance.
  Interventions: Dietary Supplement: PreMama Balance
- Placebo Drink (Placebo Comparator): Each day, the participants will take 1 packet of Placebo Drink, dissolved in one glass (8oz+) of water. Placebo Drink may be taken with or without food. Should participants present themselves with a sensitive stomach, it is recommended to take the drink with or after a meal to avoid an upset stomach. Participants will repeat this process daily for 6 months/24 weeks (study period) until the study is complete.
  At week 12 and in week 24, the participants will take a survey and a hormone test to track progress. In total there will be 3 surveys and 3 hormone tests. Additionally, participants will fill out a weekly consumption survey to track compliance.
  Interventions: Dietary Supplement: Placebo Drink

INTERVENTIONS:
Dietary Supplement: PreMama Balance — Premama Balance is a blend of the following: Vitex (Chasteberry Extract), commonly used to help regulate hormones; Antioxidants, Selenium, and Magnesium, also help support the cleansing of hormonal birth control from the liver and help strengthen the uterine lining.
  Arms: PreMama Balance
Dietary Supplement: Placebo Drink — Blended Placebo drink
  Arms: Placebo Drink

SUMMARY:
An investigation of the dietary supplement marketed as "Premama Balance" on markers of subjective wellbeing in trial participants such as common symptoms of PMS and menstrual symptoms, as well as its effects on aiding in returning to their perceived regular/normal menstrual cycle.

ELIGIBILITY:
Inclusion Criteria:

* Must be in good health (don't report any medical conditions asked in the screening questionnaire)
* Must be on hormonal birth control (containing both progesterone and estrogen) for the past 6 months & willing to stop using it to participate in the study
* Must be willing to get off of hormonal birth control for the study period
* Must be able to track their menstrual cycle
* BMI under 40
* Agree to refrain from any lifestyle changes that may affect their menstrual cycle for the duration of the study
* Willingness to adhere to the dietary supplement regimen
* Willingness to refrain from any other dietary supplements targeting the menstrual cycle and hormone control during the study period
* Is able to communicate in English
* Is willing and able to share feedback via the used technology portal
* Must provide written informed consent (ICF)

Exclusion Criteria:

* History of oncological (including ovarian cancer) or psychiatric conditions
* History of uncontrolled health conditions
* History of hysterectomy or ovariectomy
* History of diabetes & thyroid disorders
* Smoker
* More than 3 servings of alcohol a day
* Undergoing hormonal therapy of any kind
* Menopausal or peri-menopausal
* Not starting any other form of contraceptive other than condoms, abstinence, planned sexual intercourse
* Usage of any medication or herbal remedies/supplements which can affect the menstrual cycle or hormonal balance
* If currently taking allowed supplements, the dosage needs to remain the same throughout the entirety of the study

Ages: 20 Years to 42 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2022-12-30 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
Return to perceived regular/normal menstrual cycle | 6 Months
  Survey Based Assessment of changes in menstrual cycle
Changes in PMS and Menstrual Symptoms: Cramps, Bloating, Mood swings | 6 Months
  Survey-based assessment of changes in PMS and Menstrual symptoms

CONTACTS AND LOCATIONS:
Overall Officials: Susanne Mitschke, Principal Investigator — Citruslabs

IPD SHARING:
Plan to Share IPD: Undecided